CLINICAL TRIAL: NCT00284115
Title: Efficacy of a Mechanical Gait Repetitive Training Technique Compared With a Usual Rehabilitation Program on Gait Recovery in Hemiparetic Stroke Patients
Brief Title: Efficacy of a Mechanical Gait Repetitive Training Technique in Hemiparetic Stroke Patients (AVC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFSSAPS 2005/10/006; PHRC/04-02 (Other: Rennes University Hospital)
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Hemiplegia; Stroke
Keywords: Gait trainer; Hemiplegia; Rehabilitation; Stroke
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mechanical gait repetitive training (Experimental): Body weight support treadmill training technique enabling nonambulatory patients to have the repetitive practice of a gate-like movement
  Interventions: Device: Gait trainer
- Conventional rehabilitation program (Active Comparator): Physiotherapeutic conventional rehabilitation program
  Interventions: Device: Conventional rehabilitation

INTERVENTIONS:
Device: Gait trainer — Mechanical gait repetitive training
  Arms: Mechanical gait repetitive training
Device: Conventional rehabilitation — Physiotherapeutic conventional rehabilitation
  Arms: Conventional rehabilitation program

SUMMARY:
Modern concepts of gait rehabilitation after stroke favor a task-specific repetitive approach. This study aims to test the efficacy on gait recovery of a mechanized gait trainer enabling nonambulatory patients to have the repetitive practice of a gait-like movement.

DETAILED DESCRIPTION:
Modern concepts of gait rehabilitation after stroke favor a task-specific repetitive approach. The aim of the study is to test the efficacy of a body weight support treadmill training technique enabling nonambulatory patients to have the repetitive practice of a gait-like movement compared to a conventional rehabilitation program in the acute phase. Hemiparetic stroke patients will be randomly included in a 4 week rehabilitation program associating physiotherapy and gait trainer therapy or physiotherapy alone.

The primary endpoint will be the walking speed (time needed to walk 10 m) at the end of the rehabilitation program. Functional ambulatory category, walking endurance, time to self sufficient gait recovery, needing for mobility and self assistance, spasticity and economic evaluation of the two strategies will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years or more
* Hemiplegia secondary to stroke
* Interval between stroke and study inclusion of 4 month or less
* First supratentorial stroke or no motor sequelae in case of history of transient ischemic stroke
* Non ambulatory patient (Functional Ambulatory Category Stage 0 or 1)
* Being able to sit unsupported at the edge of the bed
* No severe impairment of cognition or communication
* Written informed consent

Exclusion Criteria:

* Orthopedic and/or rheumatological disease impairing mobility
* Other Neurological associated disease
* History of myocardial infarction or deep venous embolism or pulmonary embolism less than 3 months before study inclusion
* Chronic pulmonary disease
* Intolerance to stand up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Walking speed (time needed to walk 10 m) after the 4 week rehabilitation program | after 4 weeks

SECONDARY OUTCOMES:
Functional ambulatory category | Days 0, 15, 28 and 90.
Walking endurance (6 minute walk) | days 15, 28 and 90.
  distance covered in a 6 minutes confortable walk
Time to self sufficient gait recovery | Since inclusion Time
Spasticity (modified Ashworth score) | Days 0, 15, 28 and 90
Motricity index | Days 0, 15, 28 and 90
Need for mobility and self assistance (Barthel score, PMSI-SSR scores, need for physical assistance) | Days 0, 15, 28 and 90
Economic evaluation (healthcare requirements, rehabilitation unit length of stay) | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Régine Brissot, MD, Principal Investigator — CHU Rennes; Bruno Laviolle, MD, Study Chair — CHU Rennes
Locations (12):
- France (12):
  - Rééducation et Réadaptation Fonctionnelle - Hôpital Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Centre du Docteur Bouffart-Vercelli, Cervera de la Marenda
  - Centre de Rééducation de Coubert, Coubert
  - Rééducation Fonctionnelle - Hôpital Raymond Poincaré, Garches
  - Centre l'espoir, Hellemmes-Lille
  - Centre Bretegnier, Héricourt
  - Département de Médecine Physique et Réadaptation - Hôpital Jean Rebeyrol, Limoges
  - Service de Médecine Physique et Réadaptation - Hôpital de l'Archet, Nice
  - Service de Médecine Physique et Réadaptation - Centre Hospitalier Le Grau du Roi, Nîmes
  - Service de Rééducation Neuro-orthopédique - Hôpital Rothschild, Paris
  - Service de Médecine Physique et Réadaptation - Hôpital Pontchaillou, Rennes
  - Centre de l'Arche, Saint-Saturnin